CLINICAL TRIAL: NCT02896725
Title: Keratin4VLU: A Randomised Controlled Trial of Wool-derived Keratin Dressings for Venous Leg Ulcers
Brief Title: Wool-derived Keratin Dressings for Venous Leg Ulcers
Acronym: Keratin4VLU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Auckland, New Zealand (Other)
Collaborators: Health Research Council, New Zealand (Other)
Responsible Party: Principal Investigator, Andrew Jull, Associate Professor, University of Auckland, New Zealand
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Keratin4VLU; U1111-1186-5202 (Other: World Health Organisation Universal Trial Number)
Record Dates: First submitted 2016-08-29; First posted 2016-09-12 (Estimated); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Varicose Ulcer
Keywords: Venous leg ulcer; Acellular skin substitutes; Keratin dressings
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Intervention Model Description: Participants allocated to receive either keratin dressing or usual care dressing
Who Masked: Outcomes Assessor
Masking Description: Healing status for primary and secondary outcomes are adjudicated by blinded review of photographs of healed reference ulcer site or unhealed reference
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Keratin dressings (Experimental): Wool-derived keratin matrix dressing applied with each change of the compression bandage until healing
  Interventions: Device: Keratin dressings
- Usual care dressings (Active Comparator): Dressing chosen from study centres' formulary of non-medicated moist wound dressings applied with each change of the compression bandage until healing
  Interventions: Device: Usual care dressings

INTERVENTIONS:
Device: Keratin dressings — Wool-derived keratin matrix dressings applied with each change of the compression bandage until healing or the trial ends
  Arms: Keratin dressings
Device: Usual care dressings — Dressings chosen from study centres' formulary of non-medicated moist wound dressings (non-adherent dressings, hydrogel, alginate, hydrofibre or polyurethane foam dressings) applied with each change of the compression bandage until healing or the trial ends
  Arms: Usual care dressings

SUMMARY:
Venous leg ulcers (VLU) are the most common leg ulcer, can be painful, and limit work, lifestyles and activity, especially in older patients. Compression bandaging is the main treatment but there are few added treatments for patients with slow healing VLU. About 50% of patients with VLU may be slow healing. Research suggests using keratin dressings as well as using compression may help healing in patients with show healing VLU, but the current evidence is not enough to change clinical practice. The investigators will conduct a randomised controlled trial to test whether using keratin dressings is better than usual care for slow healing VLU.

DETAILED DESCRIPTION:
A pragmatic, community based, single-blind, usual care-controlled, randomised trial to determine whether keratin dressings increase the proportion of patients with venous leg ulcers healed at 24 weeks when used in addition to compression in patients with slow healing venous leg ulcers. Participants in have compression therapy (system of choice guided by patient and/or clinical preference) as delivered through district nursing services at the study centres as a background treatment. Keratin dressings will be applied when the compression bandage is changed (approximately weekly). Usual care dressings will consist of the usual formulary of moist wound dressings available at each study centre.

Participants will be district nursing service patients in five study centres in New Zealand with prevalent or incident venous leg ulcers. A venous leg ulcer will be defined as a wound on the lower leg that has remained unhealed for 4 or more weeks, appears to be primarily venous in aetiology with other causative diseases ruled out. If the participant has two or more venous leg ulcers, the largest ulcer will be the reference ulcer. A participant will be considered to have a slow healing venous leg ulcer if the ulcer area is larger than 5 cm2 and/or the ulcer has been present for more than six months.

Participants will receive up to four visits from the research nurse - visit 1 to screen for eligibility, visit 2 to consent and randomise the participant, visits 3 and 4 to collect outcome data. District nurses will continue to visit the participant (about weekly or more frequently if required) to provide routine care between research nurse visits.

Block randomisation will be used, stratified by study centre and prognostic index (ulcer size greater than 5cm2 and/or ulcer duration greater than 6 months) to ensure a balance of participants within study centres and for participants likely to be slow healers. Research nurses will input information on inclusion criteria, exclusion criteria, and relevant clinical history on consented participants via a tablet computer. The allocation will be generated after this information has been entered. Randomised participants will receive the allocated treatment until the reference ulcer heals or data collection is completed, whichever occurs sooner.

ELIGIBILITY:
Inclusion Criteria:

* Clinical indications of venous leg ulceration
* Ankle Brachial Index ≥ 0.7
* Able to tolerate compression therapy
* Ulcer area > 5cm2 and/or ulcer duration > 6 months
* Able to provide informed consent.

Exclusion Criteria:

* Hypersensitivity to wool or wool alcohols
* Venous leg ulceration with exposed tendon or bone
* Infected venous leg ulcer at trial inception (eligible after infection resolved)
* Venous leg ulcer with critical bioburden at trial inception (eligible if resolved)
* History of rheumatoid arthritis or vasculitis
* Uncontrolled diabetes
* Severe liver, heart, or renal failure
* Severe peripheral arterial disease
* Suspected or diagnosed skin malignancy
* Other threat to safe participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with complete healing of reference ulcer | 24 weeks

SECONDARY OUTCOMES:
Agreement between blinded and unblinded assessors on healing | 24 week outcome
Time to complete healing of reference ulcer | Until data collection completed two years after first participant is recruited
Change in estimated reference ulcer area | 24 weeks
  Estimated ulcer area will be derived measuring maximum width and length to determine area using formula for area of an ellipse. Such an approach is highly co-related (r=0.92) with more sophisticated measurement methods.
Change in health-related quality of life (generic) | 24 weeks
  The RAND-36 questionnaire will be used for measurement of generic health-related quality of life
Change in health-related quality of life (generic) | 24 weeks
  The EuroQuol-5D questionnaire will be used to generate utility values for cost-effectiveness modelling should that be undertaken
Change in health-related quality of life (disease-specific) | 24 weeks
  The Charing Cross Venous Ulcer Questionnaire will be used for measurement of disease-specific health-related quality of life
Incidence of adverse events | Until data collection completed two years after first participant is recruited

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Jull, RN PhD, Principal Investigator — National Institute for Health Innovation, University of Auckland
Locations (1):
- University of Auckland, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
Anonymised individual participant data may be made available on request to the Principal Investigator

REFERENCES:
- [Background] Jull A, Wadham A, Bullen C, Parag V, Waters J. Wool-derived keratin dressings versus usual care dressings for treatment of slow-healing venous leg ulceration: study protocol for a randomised controlled trial (Keratin4VLU). BMJ Open. 2018 Feb 13;8(2):e020319. doi: 10.1136/bmjopen-2017-020319. PMID 29440219
- [Derived] Jull A, Wadham A, Bullen C, Parag V, Weller C, Waters J. Wool-derived keratin dressings versus usual care dressings for treatment of slow healing venous leg ulceration: a randomised controlled trial (Keratin4VLU). BMJ Open. 2020 Jul 20;10(7):e036476. doi: 10.1136/bmjopen-2019-036476. PMID 32690743